CLINICAL TRIAL: NCT05525247
Title: A Phase 1/2, Open-label, Multicenter, Dose Escalation and Expansion Study of SLC-3010 Monotherapy and in Combination With Various Anticancer Therapies in Patients With Advanced Solid Tumors
Brief Title: A Phase 1/2, Open-label, Multicenter, Dose Escalation and Expansion Study of SLC-3010 Monotherapy and in Combination
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Selecxine (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SLC-3010-001
Record Dates: First submitted 2022-08-23; First posted 2022-09-01 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumor
Keywords: IL-2; IL-2/anti-IL-2(TCB2) conjugate; SLC-3010; Immuno-oncology
MeSH Terms: interventions — Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy (Experimental): SLC-3010 Intravenous infusion over 30 minutes on day 1 of each 21-day cycle
  Interventions: Drug: SLC-3010
- Gemcitabine combination (Experimental): SLC-3010 Intravenous infusion over 30 minutes on day 1 of each 21-day cycle
  Gemcitabine 1000 ㎎/㎡ Intravenous infusion over 30 minutes on day 1 and 8 of each 21-day cycle
  Interventions: Drug: SLC-3010; Combination Product: Gemcitabine

INTERVENTIONS:
Drug: SLC-3010 — Intravenous (IV) infusion over 30 minutes on day 1 of each 21-day cycle
Combination Product: Gemcitabine — 1000 ㎎/㎡ IV infusion over 30 minutes on day 1 and 8 of each 21-day cycle
  Arms: Gemcitabine combination

SUMMARY:
This is a Phase 1/2, open-label, multicenter, dose escalation and expansion study, evaluating the safety, tolerability, pharmacokinetic, preliminary anti-tumor activity, and effects on pharmacodynamic markers following administration of SLC-3010 as monotherapy and in combination with gemcitabine, in patients with various advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following inclusion criteria to be eligible for enrollment into the study:

1. Histologically or cytologically-documented solid tumors that are inoperable locally advanced, metastatic, or recurrent:

   * Part 1 Dose Escalation: Patients with any solid tumor who have progressed on or are intolerant to standard therapy, for which no standard therapy is available, or who decline standard therapy.
   * Part 2: Dose Expansion: Patients must have received at least one prior line of standard therapy in recurrent/metastatic setting and for whom standard life-prolonging therapies are either not available or are not qualified to receive such therapies. Additional general and tumor specific inclusion and exclusion criteria will apply.
2. Patients who have at least one measurable lesion, as defined by RECIST v1.1.
3. Adult male or female patients ≥18 years of age on day of signing the informed consent form (ICF) or follow local regulatory requirement if the legal age for consenting for study participation is more than 18 years.
4. Patients who are able and willing to provide written informed consent and are willing and able to comply with all study procedures.
5. Patients with life expectancy of ≥3 months.
6. Patients with Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
7. Patients who demonstrate adequate organ function as defined.
8. Resolution of any clinically significant toxic effects of prior therapy to Grade 0 or 1 according to the NCI CTCAE v5.0 (exception of alopecia and other AEs that are acceptable in the opinion of the Investigator and after discussion with the Medical Monitor)
9. Willingness of male and female patients of reproductive potential to observe conventional and effective birth control methods with failure rates of <1% for the duration of treatment and for 3 months (6 months for female patients administering gemcitabine) following the last dose of study treatment. This must include barrier methods such as condom or diaphragm with spermicidal gel. Women of childbearing potential (WOCBP) are defined as following menarche and who are not postmenopausal (and 2 years of nontherapy-induced amenorrhea or surgically sterile). For male patients with a nonpregnant female partner of childbearing potential and a WOCBP, 1 of the following highly effective birth control methods, with a failure rate of less than 1% per year when used consistently and correctly, is recommended:

   1. Combined estrogen and progestin containing hormonal contraception associated with inhibition of ovulation given orally, intravaginally, or transdermally
   2. Progestin-only hormonal contraception associated with inhibition of ovulation given orally, by injection, or by implant
   3. Intrauterine device
   4. Intrauterine hormone-releasing system
   5. Bilateral tubal occlusion/ligation
   6. Vasectomized partner
   7. Sexual abstinence Note: Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drug. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the patient.

   Birth control methods unacceptable for this study include the following:
   1. Periodic abstinence (calendar, symptom-thermal, or post-ovulation methods)
   2. Withdrawal (coitus interruptus)
   3. Spermicide only
   4. Lactational amenorrhea method
   5. Sperm donation is prohibited during the duration of participation on this protocol and for 90 days after the last dose of study drug
10. WOCBP must have a documented negative serum or urine pregnancy at screening within 3 calendar days before the first dose of study drug. Females who are not of childbearing potential must have documented:

    1. Postmenopausal status, defined as cessation of regular menses for at least 12 months and documented serum follicle stimulating hormone (FSH) levels that are within laboratory reference range for postmenopausal women, or
    2. Have undergone a documented hysterectomy or bilateral oophorectomy, or
    3. Have medically confirmed ovarian failure.

Exclusion Criteria:

Individuals who meet any of the following exclusion criteria will not be eligible to participate:

1. Prior history of or active malignant disease other than that being treated in this study.

   Exceptions: (i) Malignancies that were treated curatively and have not recurred within the past 2 years, or (ii) Completely resected basal cell carcinoma and squamous cell carcinoma of the skin, or (iii) Completely resected carcinoma in situ of any type.
2. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/ or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study drug. Note: patients with an incidental finding of an isolated lesion <1 cm in diameter may be eligible if the lesion does not require treatment per investigator judgment. Eligible patients must be neurologically asymptomatic and without corticosteroids treatment for at least 2 weeks prior to start of first dose of study treatment.
3. Diagnosis of immunodeficiency or receiving chronic systemic steroid therapy, or any immunosuppressive therapy within 7 days prior to first dose of study drug. Topical (<class III), inhaled, nasal, and ophthalmic steroids are allowed.
4. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
5. History of Grade 3 or higher immune mediated AEs that were considered drug related to prior immunotherapy (e.g., checkpoint inhibitors, co-stimulatory agents).
6. Infection with HIV-1 or HIV-2. Active hepatitis B (hepatitis B virus [HBV] surface antigen positive), hepatitis C (hepatitis C virus [HCV] antibody positive, confirmed by HCV ribonucleic acid). Patients with prior history of HBV are eligible if quantitative polymerase chain reaction (PCR) for HBV DNA is negative. Patients with HCV with undetectable virus after treatment, and those who have minimal viral load (<20 IU/ml) at screening and who are being treated with HCV therapy during the full study period are eligible.
7. Has an active infection requiring systemic therapy
8. Has significant cardiovascular disease, such as:

   1. QT interval corrected for heart rate using Fridericia's formula > 480 msec at screening
   2. History of myocardial infarction, acute coronary syndrome or coronary angioplasty/stenting/bypass grafting within the last 6 months
   3. Congestive heart failure (CHF) New York Heart Association (NYHA) Class II-IV or history of CHF NYHA class III or IV
9. Patients exhibiting significant respiratory symptoms, those with suspected or known serious or severe respiratory conditions and those requiring supplemental oxygen at screening.
10. Receipt of any type of systemic anticancer therapy (including investigational therapy) within 3 weeks before the first dose of study drug or 5 times elimination half-life of drug, if known, has passed whatever is shorter.
11. Is currently participating in or has participated in an interventional clinical trial with last dose of the investigational compound or device within 3 weeks of the first dose of treatment in this current trial. Patients who are in survival follow up can be enrolled if the last dose was 3 weeks earlier.
12. Radiation within 2 weeks before first dose of study treatment. Patients with clinically relevant ongoing complications from prior RT are not eligible.
13. Major surgery within 2 weeks prior to study drug administration; patients must have recovered adequately from toxicity and/ or complications per investigator discretion.
14. Receipt of any live vaccines within 4 weeks prior to first dose of study drug.
15. Receipt of non-live COVID-19 vaccine within 7 days prior to DLT evaluation because vaccine related toxicities could interfere safety assessment.
16. Any prior treatment with IL-2 based drug.
17. Has a known hypersensitivity to the components of the study therapy or its analogs.
18. Has a history or current evidence of any condition therapy, lab abnormality or other circumstance that might expose the patient to risk by participating in the trial, confound the results of the trial, or interfere with the patient's participation for the full duration of the trial.
19. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
20. For women only: pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of DLTs | 30 days after last dose
  Number of participants with DLTs of SLC-3010 treatment

CONTACTS AND LOCATIONS:
Locations (9):
- United States (3):
  - Selecxine Investigator site, Sarasota, Florida
  - Selecxine Investigator site, Detroit, Michigan
  - Selecxine Investigator site, Oklahoma City, Oklahoma
- Australia (2):
  - Selecxine Investigator site, Waratah, New South Wales
  - Selecxine Investigator site, Brentwood, Perth
- South Korea (4):
  - Selecxine Investigator site, Seoul, Jongno-gu
  - Selecxine Investigator site, Seoul, Seodaemun-gu
  - Selecxine Investigator site, Gyeonggi-do, Seongnam-si
  - Selecxine Investigator site, Seoul, Songpa-gu

IPD SHARING:
Plan to Share IPD: No